CLINICAL TRIAL: NCT03560700
Title: The Effect of a Lactobacillus Probiotic Strain on Eradication of Vancomycin Resistant Enterococcus Faecium (VRE) in Non-symptomatic VRE-carriers - a Multicenter, Randomized, Placebo-controlled, Parallel-group Study With 4 Weeks Intervention
Brief Title: Probiotic Efficacy in VRE Eradication
Acronym: PROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Chr Hansen (Industry)
Responsible Party: Principal Investigator, Andreas Munk Petersen, Md, Phd, Consultant, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-18011991
Record Dates: First submitted 2018-05-24; First posted 2018-06-18 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: VRE Colonization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lactobacillus probiotic strain (Experimental): 60 billion CFU/day
  Interventions: Dietary Supplement: lactobacillus probiotic strain
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: lactobacillus probiotic strain — Approved Dietary supplement
  Arms: lactobacillus probiotic strain
Other: placebo — placebo comparator
  Arms: placebo

SUMMARY:
This study will evaluate the efficacy of a probiotic lactobacillus strain in eradicating VRE in non-symptomatic carriers after 4 weeks of treatment. It will also evaluate the long-term efficacy after 8,16 and 24 weeks.

DETAILED DESCRIPTION:
With the increased number of Vancomycin-Resistant Enterococcus faecium (VRE) infected/colonized people it is evident that new treatment options are needed to reduce the number of VRE cases. One such option could be to use probiotics. We hypothesize that treatment with a probiotic lactobacillus strain can reduce the number of VRE carriers significantly. The aim is to investigate if this strain can eradicate VRE in non-symptomatic VRE-carriers measured as the number of subjects without VRE colonization at week 4.

This is a multi-center, randomized, double-blind, placebo-controlled parallel-group trial in non-symptomatic VRE-carriers.

The Trial consists of a 4 weeks intervention period followed by a 20-week follow-up period.

After patients have been confirmed as carriers of VRE, the subjects are randomized to 4 weeks' treatment with a lactobacillus probiotic strain (60 billion CFU per day) or to placebo. Subjects' VRE carrier-state is assessed at weeks 4, 8, 16 and 24, by an in-house PCR analysis. Stool samples are collected before intervention (baseline) and at week 4, 8, 16 and week 24.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with VRE colonization (positive faecal swab)
* Subjects over 18 years of age
* Provided voluntary written informed consent

Exclusion Criteria:

* Symptomatic VRE infection
* Serious immunodeficiency
* Pancreatitis
* Planned or recent intraabdominal operation within a time window of14 days)
* Parenteral nutrition
* Antibiotic treatment for VRE one month prior to inclusion
* Terminal disease with expected survival time < 3 month
* Probiotic consumption within two weeks prior enrollment
* Pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with cleared VRE colonization at week 4 | 4 weeks
  Fecal sample diagnosed by pcr and detection of the vanA gene

SECONDARY OUTCOMES:
Clearance of VRE colonization at week 8, 16 and 24 respectively | 8, 16 and 24 weeks
  Fecal sample diagnosed by pcr and detection of the vanA gene
Number of VRE infections (isolation from non-intestinal foci) | 24 weeks
Changes in fecal microbiota composition | 24 weeks
Colonization with probiotic lactobacillus strain | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Copenhagen University, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rubin IMC, Mollerup S, Broholm C, Knudsen SB, Baker A, Helms M, Holm MKA, Kallemose T, Westh H, Dahl Knudsen J, Pinholt M, Petersen AM. No Effect of Lactobacillus rhamnosus GG on Eradication of Colonization by Vancomycin-Resistant Enterococcus faecium or Microbiome Diversity in Hospitalized Adult Patients. Microbiol Spectr. 2022 Jun 29;10(3):e0234821. doi: 10.1128/spectrum.02348-21. Epub 2022 Apr 27. PMID 35475684